CLINICAL TRIAL: NCT06005610
Title: Giving Standardized Estradiol Therapy In Transgender Women to Research Interactions With HIV Therapy
Brief Title: Estradiol Therapy In Transgender Women to Research Interactions With HIV Therapy
Acronym: GET IT RIgHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5403; 38806 (Other: DAIDS-ES ID)
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-06

CONDITIONS: HIV I Infection
Keywords: HIV; Transgender women; Estradiol; ART; Drug interactions
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: BIC-treated (Experimental): Participants taking bictegravir (BIC) + tenofovir alafenamide (TAF) + emtricitabine (FTC)
  Interventions: Drug: Estradiol
- Group 2: DTG-treated (Experimental): Participants taking dolutegravir (DTG) once daily + tenofovir disoproxil fumarate (TDF) + (FTC or lamivudine [3TC])
  Interventions: Drug: Estradiol
- Group 3: Boosted DRV-treated (Experimental): Participants taking any regimen containing darunavir plus cobicistat (DRV/c)
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — Oral 17-β estradiol 2 mg once daily will be initiated at study entry. At weeks 4, 12, 24, and 36, study clinicians may titrate 17-β estradiol in 2 mg increments to achieve the desired participant goals and target hormone concentrations, as measured locally at each visit.

SUMMARY:
Transgender women (TW) are a key population and priority for HIV treatment. More research is needed to develop evidence-based clinical guidance when it comes to choosing antiretroviral treatment (ART) regimens for TW on feminizing hormonal therapy (FHT). Concerns about ART interacting with FHT and decreasing its effectiveness can lead to decreased ART adherence and increased viral loads.

The GET IT RiGHT trial aims to address concerns about drug-drug interactions (DDIs) between ART and FHT while providing access to hormonal therapy to TW living with HIV. Data suggest that access to FHT improves adherence to HIV treatment and decreases treatment interruptions.

This is an open-label, non-randomized, 3-group trial of adult TW and other individuals identifying as female or transfeminine but with male sex assigned at birth living with HIV. Participants will be on ART at entry and receive study-supplied 17-β estradiol for FHT for 48 weeks.

The primary objectives of the study are to 1) assess whether TW continue to achieve therapeutic concentrations of ART while receiving FHT for 48 weeks and 2) assess whether serum estradiol concentrations on FHT (across a range of estradiol doses) vary between boosted and un-boosted ART regimens.

DETAILED DESCRIPTION:
A5403 is a phase IIb, 48-week, open-label, non-randomized, 3-group trial, of 90 adult (≥18 years) transgender women and other individuals identifying as female or transfeminine but with male sex assigned at birth (TW) living with HIV on suppressive antiretroviral therapy (ART) and not currently on FHT. The trial will target at least 50% enrollment of participants identifying as non-white or Latine.

The trial consists of three groups, a BIC-treated group (BIC/TAF/FTC; n=30) (Group 1), a DTG-treated group (DTG/TDF/FTC or 3TC; n=30) (Group 2), and a boosted DRV-treated group (DRV/c; n=30) (Group 3), for a total of 90 participants.

All participants will continue on ART (not provided by the trial) and receive study-supplied 17-β estradiol for weeks 0-48. At entry, participants will be assigned to one of the three analysis groups based on their current ART regimen. Participants on other ART regimens at screening who are willing to switch to one of the regimens above, may also be enrolled.

All participants will receive study supplied 17-β estradiol for weeks 0-48. Oral 17-β estradiol 2 mg once daily will be initiated at study entry. At weeks 4, 12, 24, and 36, study clinicians may titrate 17-β estradiol in 2 mg increments as described in the protocol.

Intensive PK subgroup (n=15 per ART group): At entry (week 0), an 8-hour intensive PK sampling will assess ART exposure prior to FHT initiation. At week 24, intensive sampling will be repeated to assess 17-β estradiol and ART exposure. A final intensive PK visit will occur at week 48 to assess 17-β estradiol and ART exposure at the maximal FHT dosing achieved during the study period.

Sparse PK sampling: all participants not participating in an intensive PK sampling visit on the same day will have timed, sparse PK sampling collected at each visit to characterize the trough plasma (BIC, DTG, and DRV) and intracellular ART (TFV-DP, FTC-TP, 3TC-TP) concentrations to evaluate the relationship of ART PK exposure across a range of 17-β estradiol doses.

FHT satisfaction and acceptability:

To measure acceptability, participants will be asked to self-report the degree to which they find the intervention appropriate and useful using Likert-type agreement scales at three study time points: entry, 24 weeks, and 48 weeks. To measure satisfaction, the 12-question Transgender Congruence Scale (TCS) will be used, which will assess associations between gender-affirming treatments, perceived gender congruence, and satisfaction at three study time points: entry, 24 weeks, and 48 weeks. In addition, brief, 20-minute, semi-structured interviews will be conducted with 30 purposively sampled participants across English- or Spanish-speaking sites to provide an opportunity for more in-depth (open-ended) feedback on intervention satisfaction and acceptability at three time points: entry, 24 weeks, and 48 weeks.

Other assessments throughout the study include: anthropometric measurements (including weight, height, minimum waist circumference, and maximum hip circumference), routine chemistry and hematology labs, HIV-1 RNA, CD4+ and CD8+ T cell counts and percentages, lipids, glucose and insulin, non-estradiol hormone concentrations, stored PBMC, plasma, and serum, and ART and FHT adherence assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Documentation of HIV-1 status.
3. Assigned male sex at birth and identifies as a TW, female or transfeminine person.
4. On ART for at least 24 weeks prior to study entry. Regimen changes within the 24 weeks prior to study entry are acceptable, but candidates must have been on a stable regimen for at least 28 days prior to study entry.
5. On BIC/FTC/TAF, DTG/TDF/FTC or 3TC, or DRV/c-containing ART for at least 28 days prior to study entry (single tablet regimen not required), and with no plans to change ART regimen over the study duration of 48 weeks.
6. Desire to initiate or restart FHT, regardless of orchiectomy status.
7. HIV-1 RNA <200 copies/mL at screening.
8. HIV-1 RNA <400 copies/mL available through routine clinical care between 24 and 96 weeks prior to study entry and while on ART. The HIV-1 RNA must be the most recent value obtained between 24 and 96 weeks prior to study entry.
9. The following laboratory values obtained within 60 days prior to study entry

   * Hemoglobin ≥9.0 g/dL
   * Platelet count ≥75,000/mm3
   * Estimated Glomerular Filtration Rate (eGFR) ≥30 mL/min/1.73m2 if on or switching to TAF, ≥50 mL/min/1.73m2 if on or switching to TDF without cobicistat, or ≥70 mL/min/1.73m2 if on or switching to TDF in combination with cobicistat, calculated using the CKD-Epi equation
   * Aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), and alkaline phosphatase are within normal range per local laboratory range
   * Prolactin <25 ng/dL
10. Serum estradiol level <75 pg/mL within 60 days prior to study entry.
11. Willingness to avoid the use of prescribed, non-study provided FHT and non-prescribed FHT during the study period, and no planned use of prescribed or non-prescribed anti-androgens for the first 24 weeks of the study.
12. Ability and willingness of participant to provide informed consent and ability and willingness of participant to undergo study procedures.

Exclusion Criteria:

1. Known clotting disorders, active deep vein thrombosis (DVT), pulmonary embolism (PE), or history of these conditions, active arterial thromboembolic disease (e.g., stroke, myocardial infarction), or history of these conditions.
2. Known liver impairment or disease.
3. History of chronic hepatitis B virus (HBV) infection or active HBV infection.
4. History of current active hepatitis C virus (HCV) infection.
5. Prohibited medication use (including drugs with known or expected DDIs with FHT or ART) at time of study entry.
6. Receipt of any estrogen therapy within 14 days prior to study entry for persons on oral FHT, or within 30 days prior to entry for persons on injectable FHT.
7. Known HIV-1 resistance mutations that would preclude remaining on current ART or a switch to a study regimen, in the opinion of the site investigator.
8. Personal history of breast cancer. or known personal history of breast cancer (BRCA) gene.
9. Known or a history of testicular cancer.
10. Known or a history of gall bladder disease.
11. Known or suspected pituitary adenoma.
12. Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
13. Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
14. Suicidal ideation in the past 30 days or suicide attempt in the past 90 days, as reported on the Columbia-Suicide Severity Rating Scale (C-SSRS).
15. Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry. Stable (in the opinion of the site investigator) treatments for chronic comorbidities are allowed.
16. Presence of any other medical condition that would preclude FHT administration for safety reasons, in the opinion of the site investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned male sex at birth and identifies as a TW, female or transfeminine person.
Enrollment: 93 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Ratio of ART Analytes BIC, DTG, and DRV trough concentrations (Ctrough) in plasma at each received dose of oral 17-β estradiol | Study Entry and Weeks 4, 12, 24, 36, and 48
  Log-transformed trough concentrations (Ctrough) in ng/mL of the analytes BIC, DTG, and DRV from plasma samples collected 22-26 hours post ART dose, measured over 48 weeks.
Percentage of Participants with ART Analyte trough concentration (Ctrough) above drug-specific threshold | Study Entry and Weeks 4, 12, 24, 36, and 48
  Trough concentration of the analytes BIC, DTG, and DRV in plasma at each received dose of 17-β estradiol summarized at the participant level as indicator of concentration being above drug-specific threshold.
Trough serum total estradiol assessed at each received dose of oral 17-β estradiol as quantified via batch testing at central lab. | Study Entry and Weeks 4, 12, 24, 36, and 48
  Trough concentrations of Total 17-β estradiol in ng/mL from serum samples collected 22-26 hours post 17-β estradiol dose. Results < Lower Limit of Quantification (LLoQ) at entry will be imputed as 0 ng/mL at one-half the LLoQ value at visits post-entry.

SECONDARY OUTCOMES:
Trough concentrations of TFV-DP, FTC-TP, and 3TC-TP in non-viable PBMCs at each received dose of oral 17-β estradiol | Study Entry and Weeks 4, 12, 24, 36 and 48
  Intra-person geometric ratios of trough ART concentration at each received estradiol dose relative to pre-FHT (i.e., baseline).
Percentage of Participants with TFV-DP, FTC-TP, and 3TC-TP trough concentration above drug-specific threshold | Study Entry and Weeks 4, 12, 24, 36 and 48
  Trough concentration of the analytes TFV-DP, FTC-TP, and 3TC-TP in non-viable PBMCs at each received dose of 17-β estradiol summarized at the participant level as indicator of concentration being above drug-specific externally defined threshold.
Percentage of participants with an occurrence of any reportable adverse event related to 17-β estradiol | Study entry to Week 48
  The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017, and the DAIDS EAE Manual Version 2.0 will be used.
Percentage of participants with an occurrence of SAEs as defined by International Conference on Harmonization (ICH) and new events of CAD/CVD, cancer, DM/pre-DM, and vascular event | Study entry to Week 48
  Post-entry and while on study treatment, all signs (including an abnormal laboratory finding), symptoms, or diagnoses new in onset or aggravated in severity or frequency from the baseline condition, indicated as related to 17-β estradiol by the site (or the CMC if adjudication differs from that of the site investigator).
Percentage of participants with serum total testosterone < 50 ng/dL at each received dose of oral 17-β estradiol | Study entry and Weeks 4, 12, 24, 36, 48
  Results < LLoQ will be considered to be <50 ng/dL. If multiple observations are available at the same estradiol dose, the last testosterone concentration (based on calendar time) taken will be used.
Percentage of participants with virologic suppression of HIV | Study entry and weeks 12, 24, 36, and 48
  Virologic suppression of HIV is defined as plasma HIV-1 viral load <50 copies/mL
Absolute changes in overall transgender congruence score | Study entry and weeks 24, and 48
  The overall transgender congruence score is calculated from participant response to the 12-question Transgender Congruence Scale (TCS). Participants rate each item on a 5-point Likert-type scale (i.e., 1 = strongly disagree, 2 = somewhat disagree, 3 = neither agree nor disagree, 4 = somewhat agree, 5 = strongly agree). Questions 'The way my body currently looks does not represent my gender identity.', 'I do not feel that my appearance reflects my gender identity.', and 'I am not proud of my gender identity.' are reversed scored. The overall score is the average of the response to the 12 questions, with higher scores indicating a higher level of congruence. Positive changes from baseline indicate improvement in transgender congruence.
Area under the curve over 8 hours (AUC 0-8h) of 17-β estradiol | Study entry and Weeks 24, and 48
  From pre-dose, 1, 2, 3, 4, 6, and 8 hours post dosing at entry and weeks 24 and 48.
  The AUC will use the linear up/log down version of the trapezoidal rule in non-compartmental analysis using Phoenix WinNonLin (Certara®). This version of the trapezoidal rule uses linear interpolation between untransformed data up to Cmax, and between log-transformed data from Cmax through Clast.
Percent change in weight | Study entry and weeks 12, 24, 36, and 48
  Calculated by dividing weight at later time point minus weight at study entry by weight at study entry.
Percent change in BMI | Study entry and weeks 12, 24, 36, and 48
  Calculated by dividing BMI at later time point minus BMI at study entry by BMI at study entry.
Absolute change in minimum waist circumference | Study entry and weeks 12, 24, 36, and 48
  Calculated as waist circumference at later time point minus waist circumference at study entry.
Absolute change in maximum hip circumference | Study entry and weeks 12, 24, 36, and 48
  Calculated as maximum hip circumference at later time point minus maximum hip circumference at study entry.
Absolute change in waist-hip ratio measured | Study entry and weeks 12, 24, 36, and 48
  Calculated as waist-hip ratio at later time point minus waist-hip ratio at study entry.
Absolute changes in fasting lipids | Study entry and weeks 12, 24, and 48
  Calculated as fasting lipids at later time point minus fasting lipids at study entry.
Absolute changes in glucose sensitivity | Study entry and weeks 12, 24, 36, and 48
  Calculated as glucose sensitivity at later time point minus glucose sensitivity at study entry.
Absolute changes in insulin sensitivity | Study entry and weeks 12, 24, 36, and 48
  Calculated as insulin sensitivity at later time point minus insulin sensitivity at study entry. Insulin will be measured from stored samples. Insulin sensitivity will be calculated as: HOMA-IR = (fasting glucose in mmol/L * fasting insulin in µU/L) /22.5.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan E. Lake, MD, MSc, Study Chair — Houston AIDS Research Team CRS; Kimberly K. Scarsi, PharmD, MS, FCCP, Study Chair — University of Nebraska; Jorge A. Gallardo-Cartagena, MD, Study Chair — Barranco CRS
Locations (18):
- United States (14):
  - UCSD Antiviral Research Center CRS (701), San Diego, California
  - University of California, San Francisco HIV/AIDS CRS (801), San Francisco, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Whitman-Walker Institute, Inc. CRS (31791), Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS (5802), Atlanta, Georgia
  - Johns Hopkins University CRS (201), Baltimore, Maryland
  - Washington University Therapeutics (WT) CRS (2101), St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS (31786), Newark, New Jersey
  - Weill Cornell Uptown CRS (site 7803), New York, New York
  - Chapel Hill CRS (3201), Chapel Hill, North Carolina
  - Greensboro CRS (3203), Greensboro, North Carolina
  - Case CRS (2501), Cleveland, Ohio
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - Houston AIDS Research Team CRS (31473), Houston, Texas
- Nutrición-Mexico CRS (32078), Mexico City, Tlalpan, Mexico
- Barranco CRS (11301), Lima, Peru
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS (31802), Bangkok, Patumwan
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS (31784), Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.